CLINICAL TRIAL: NCT02693951
Title: Efficiency and Safety of Prophylactic Use of Antibiotics in Endoscopic Injection of Tissue Adhesive in Gastric Varices: A Randomized Controlled Trial
Brief Title: Efficiency and Safety of Prophylactic Use of Antibiotics in Endoscopic Injection of Tissue Adhesive in Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSY-LCF-2016
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Varices; Cirrhosis
Keywords: gastric varices; endoscopic injection of tissue adhesive
MeSH Terms: conditions — Esophageal and Gastric Varices; Fibrosis | interventions — Cefotiam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the prophylactic use of antibiotics group (Experimental): Half an hour before endoscopic treatment, cefotiam 2.0g intravenous
  Interventions: Drug: Cefotiam
- Control (No Intervention): Routine endoscopic examination and treatment. Antibiotics are not used before endoscopic treatment

INTERVENTIONS:
Drug: Cefotiam — Prophylactic use of antibiotics group: Half an hour before endoscopic treatment, cefotiam 2.0g intravenous
  Other Names: HaiTiShu
  Arms: the prophylactic use of antibiotics group

SUMMARY:
The purpose of the study is to assess the efficiency and safety of prophylactic use of antibiotics in endoscopic injection of tissue adhesive in gastric varices.

DETAILED DESCRIPTION:
At present, there is still a controversy about the application of antibiotics in the treatment of patients with non acute hemorrhage of esophageal varices. This study is a randomized controlled trial. Patients randomly enter two treatment groups:

1. the prophylactic use of antibiotics group

   and
2. the non-prophylactic use of antibiotics group

Treatment allocation is by block randomization with an equal number for both groups. The incidence of infection after endoscopic treatment will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the purpose and risks of the study and informed consent to participate in the study;
* age between 18-75 years old;
* Diagnosis of esophageal gastric varices by gastroscopy
* Preparation of endoscopic injection of tissue adhesive

Exclusion Criteria:

* No esophageal gastric varices bleeding history;
* Esophageal varices or gastric varices which temporarily won't be treated by endoscopic therapy;
* The cefotiam contraindications: such as allergies, pregnancy etc;
* Patients with the other malignant tumor except liver cancer;
* The preoperative diagnosis of infection;
* The large amount of ascites;
* The acute bleeding period (< 5 days);
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of infection after endoscopic treatment | 1 week
  Patients will receive body temperature, blood routine, inflammatory markers examination before and after endoscopic treatment.

SECONDARY OUTCOMES:
Rebleeding rate | 2 months
  Patients will receive an endoscopic examination after patients have been followed up for 2 months.
Mortality rate | 2 months
  The investigators observe the mortality events during 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China